CLINICAL TRIAL: NCT07041775
Title: MINT Conditioning to Improve Post-stroke Gait
Brief Title: MINT Conditioning to Improve Gait
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Marc Slutzky, Professor of Neurology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00221627; R01HD113270 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Stroke Gait Rehabilitation
Keywords: Stroke rehabilitation; Leg impairment; Walking; Rehabilitation gaming; Muscle biofeedback; Myoelectric interface
MeSH Terms: conditions — Stroke | interventions — Neurological Rehabilitation; SPEN protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINT group (Experimental): MINT training of two leg muscles
  Interventions: Other: myoelectric interface for neurorehabilitation (MINT) conditioning
- Sham group (Sham Comparator): one muscle feedback
  Interventions: Other: One muscle myoelectric feedback

INTERVENTIONS:
Other: myoelectric interface for neurorehabilitation (MINT) conditioning — Myoelectric interface for neurorehabilitation (MINT) conditioning involves training to reduce abnormal co-activation of limb muscles to improve movement.
  Arms: MINT group
Other: One muscle myoelectric feedback — Training to control muscle activity in one muscle only.
  Arms: Sham group

SUMMARY:
This study will test the ability of myoelectric interface for neurorehabilitation (MINT) training to improve walking function.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment is 18 to 85
* Leg impairment from unilateral stroke at least 6 months prior to screening
* Severe to moderate gait impairment (ambulatory with a maximum walking speed of 0.8 m/s, i.e., half of normal speed)
* Able to stand without assistance
* Clinically observable gait asymmetry
* Abnormal co-activation between adductor magnus and rectus femoris (R greater than or equal to 0.5)

Exclusion Criteria:

* Cognitive impairment with at least moderately impaired attention on digit-span test, or unable to follow instructions of the MINT task
* Visual impairment (such as hemianopia) preventing sufficient perception of the screen to play the games
* Anesthesia or severe neglect in the affected leg, or visual hemineglect (score of 2 on the NIH Stroke Scale Extinction and Inattention subtest) that impairs ability to play the games
* Participation in another study on the affected leg, or any pharmacological study, within 6 weeks of enrollment
* Inability to understand or follow commands in English due to aphasia or other reason that makes it impossible to perform the training
* Diffuse or multifocal infarcts
* Substantial leg or other pain preventing participation for 60 minutes a day
* Spasticity treatment (pharmacological or Botox) on the affected leg within past 3 months
* Contraindication to MRI (metal implants, pacemakers)
* History of epilepsy in adulthood
* Skull abnormalities or fractures near the motor cortex
* Severe osteoporosis causing hip or other fractures
* History of multiple falls within the last year, use of walker for balance, or falling during stance while in the lab in the first session.
* Contracture limiting the range of motion of the leg
* Current pregnancy
* Absence of MEP using TMS (lack of intact corticospinal tract)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
10-m walk test | Baseline and 4 weeks
  The 10-m walk test measures gait speed

SECONDARY OUTCOMES:
6-min walk test | Baseline and week 4
  The 6-min walk test measures the distance subjects can walk in 6 min. It measures endurance.
10-m walk test | Baseline and week 8
  The 10-m walk test measures gait speed
6-min walk test | Baseline and week 8
  The 6-min walk test measures the distance subjects can walk in 6 min. It measures endurance.
MINT performance | each training session
  The mean weighted time-to-target over trials.
Target muscle co-activation | Baseline and weeks 4 and 8
  The co-activation (correlation) between the targeted muscles daily during training and in the lab sessions during the evaluation times.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Slutzky, MD, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data and metadata will be shared in the Data Archive for the BRAIN Initiative (DABI) database. Clinical functional outcomes, gait kinematics, and analyzed EMG (co-activation), will be uploaded and shared upon publication.
Supporting Information: Analytic Code
Time Frame: IPD and associated analytic code will be made available upon publication of research results and will remain available for the duration of the funded project.